CLINICAL TRIAL: NCT04138823
Title: An Open Label, Phase I Study of BI 891065 Monotherapy and Combination Therapy of BI 891065 and BI 754091 in Asian Patients With Advanced Solid Tumours
Brief Title: A Study to Test Different Doses of BI 891065 Alone and in Combination With BI 754091 in Asian Patients With Different Types of Advanced Cancer (Solid Tumours)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1379-0006
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: 100 mg BI 891065 QD (Experimental)
  Interventions: Drug: BI 891065
- Part A: 200 mg BI 891065 QD (Experimental)
  Interventions: Drug: BI 891065
- Part A: 200 mg BI 891065 BID (Experimental)
  Interventions: Drug: BI 891065

INTERVENTIONS:
Drug: BI 891065 — film-coated tablets

SUMMARY:
The primary objective of this trial is:

Part A

- To determine the Maximum tolerated dose (MTD) and/or the recommended dose (RD) of BI 891065 monotherapy for further development in Asian patients with advanced solid tumours

Part B

- To determine the MTD and/or the RD of BI 891065 in combination with a fixed dose of BI 754091 at 240 mg for further development in Asian patients with advanced solid tumours

The secondary objectives are:

Part A

- To document the safety and tolerability, and characterise pharmacokinetics (PK) of BI 891065 as monotherapy in Asian patients with advanced solid tumours

Part B

- To document the safety and tolerability, and characterise PK of the combination therapy of BI 891065 and BI 754091 in Asian patients with advanced solid tumours

ELIGIBILITY:
Inclusion criteria:

* Of legal age (according to local legislation) at screening. No upper limit.
* Signed and dated written informed consent in accordance with International Council on Harmonisation (ICH) Good Clinical Practice (GCP) and local legislation prior to admission to the trial.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, starting with the screening visit and through 6 months after the last dose of study treatment. A list of contraception methods meeting these criteria is provided in the patient information. The requirement of contraception does not apply to women of no childbearing potential and men not able to father a child, but they must have an evidence of such at screening.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 1
* Patients with a confirmed diagnosis of advanced, unresectable and/or metastatic solid tumours, who have failed standard treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to standard therapies.
* Presence of at least one measureable lesion according to Response Evaluation Criteria In Solid Tumours (RECIST) 1.1.
* Life expectancy of at least 12 weeks after the start of the treatment according to the Investigator's judgement
* For Part B: Patients must have at least 1 tumour lesion amenable to biopsy, and must be willing to undergo a biopsy prior to first treatment and after 3 weeks while on therapy.
* For Part B: Patients with following cancer types: bladder, colon, breast, NSCLC, ovarian, pancreatic, renal, esophagogastric, sarcoma, prostate, and melanoma

Exclusion criteria:

* Major surgeries (major according to the Investigator's assessment) performed within 12 weeks prior to the first administration or planned within 12 months after screening (e.g., hip replacement), or moderate surgeries (moderate according to the Investigator's assessment) performed within 4 weeks prior to the first administration.
* Presence of active invasive cancers other than the one treated in this trial within 5 years prior to screening, except for appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumours considered cured by local treatment
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Previous administration of BI 891065 or other Second Mitochondrial Activator of Caspases (SMAC) mimetic/IAP inhibitor
* Patients who have been treated with any other anticancer drug or investigational drug, within 4 weeks or within 5 half-life periods (whichever is shorter) prior to first administration of BI 891065
* Persistent toxicity from previous treatments that has not resolved to ≤ Grade 1 (except for alopecia and Grade 2 neuropathy due to previous treatments)
* Active, known or suspected autoimmune disease except vitiligo or resolved asthma/atopy
* (Part B only) Patients removed from previous anti-Programmed-cell-death-protein-1 (PD-1) or anti-Programmed-cell-death ligand-1 (PD-L1) therapy because of a severe immune-related adverse event (irAE)
* History (including current) of interstitial lung disease or pneumonitis within 5 years
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTcF) >480 msec
  * Any clinically important abnormalities (as assessed by the investigator) in rhythm, conduction, or morphology of resting Electrocardiograms (ECGs), e.g., complete left bundle branch block, third degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication with known or possible risk of QT interval prolongation
  * Patients with an ejection fraction (EF) of either <50% or less than the lower limit of normal of the institutional standard will be excluded, whichever is lower. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF, will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram [ECHO], multi-gated acquisition scan [MUGA]). A historic measurement of EF no older than 6 months prior to first administration of study drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both
* Inadequate organ function or bone marrow reserve as demonstrated by the following laboratory values:

  * Absolute neutrophil count (ANC) <1.5 x 109/L (<1500/mm^3)
  * Platelet count <100 x 10^9/L (<100,000/mm^3)
  * Haemoglobin <9.0 g/dL
* Alanine transaminase (ALT) >3 times the upper limit of normal (ULN) if no demonstrable liver lesion(s) (primary or metastases) or >5 times ULN in the presence of liver lesion(s)

  * Aspartate aminotransferase (AST) >3 times the ULN if no demonstrable liver lesion(s) or >5 times ULN in the presence of liver lesion(s)
  * Total bilirubin >1.5 times ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin >3.0 times ULN or direct bilirubin >1.5 times ULN
  * Serum creatinine > 1.5 x ULN (measured by enzymatic assay, Isotope dilution mass spectroscopy [IDMS] standardised Jaffe assay, or non-IDMS Jaffe assay). If serum creatinine is > 1.5 x ULN, patient is eligible if concurrent estimated glomerular filtration rate (eGFR) is ≥ 30 mL/min/1.73m^3 (measured or calculated by Chronic Kidney Disease Epidemiology [CKD-EPI] formula)
* Human immunodeficiency virus (HIV) infection. Test results obtained in routine diagnostics are acceptable if done within 6 months before the informed consent date.
* Any of the following laboratory evidence of hepatitis virus infection.

  * Positive results of hepatitis B surface (HBs) antigen
  * Presence of hepatitis B core (HBc) antibody together with hepatitis virus B (HBV) Deoxyribonucleic acid (DNA)
  * Presence of hepatitis virus C (HCV) antibody together with HCV Ribonucleic acid (RNA) In Part A, test results obtained in routine clinical practice are acceptable if done within 6 months before the informed consent date.
* Known relevant hypersensitivity to the trial drugs or their excipients based on the investigator's assessment
* Serious concomitant disease or medical condition affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as cardiac, neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the Investigator would make the patient inappropriate for entry into the trial.
* Chronic alcohol or drug abuse or any condition that, in the Investigator's opinion, makes them an unreliable trial patients, unlikely to complete the trial, or unable to comply with the protocol procedures
* Women who are pregnant, nursing, or who plan to become pregnant during the trial. Women who are nursing can be enrolled if they stop nursing. In this case, the patient cannot resume nursing even after discontinuation of study treatment.
* Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may participate provided they are stable (i.e., without evidence of Progressive disease (PD) by imaging for at least 4 weeks prior to the first dose of trial treatment, and any neurologic symptoms have returned to baseline), and there is no evidence of new or enlarging brain metastases
* Patients with known leptomeningeal disease
* Patients receiving systemic treatment with any immunosuppressive medication within 1 week prior to treatment start (steroids of max. 10 mg/day prednisolone equivalent per day are allowed, topical and inhaled steroids are not considered as immunosuppressive).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Hospital, Tokyo, Chuo-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Patel MR, Hamilton EP, George B, Kretschmar G, Harada A, Graeser R, Eleftheraki A, Tachibana Y, Yamamoto N. The Second Mitochondria-Derived Activator of Caspases Mimetic BI 891065 in Patients With Advanced Solid Tumors: Results From Two Phase I Studies. Cancer Med. 2025 Dec;14(24):e71451. doi: 10.1002/cam4.71451. PMID 41408891
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was designed as a Phase I, open-label, non-randomised, uncontrolled, multicentre trial to determine the maximum tolerated dose (MTD) or recommended dose of BI 891065, administered as single agent in Part A and in combination with 240 mg of BI 754091 (ezabenlimab) in Part B. After completion of Part A of the trial, Part B of the trial was cancelled as a whole.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Part A: 100 mg BI 891065 QD: Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered once daily (QD) orally 100 milligrams (mg) of BI 891065, composed of two 50 mg film-coated tablets, with 240 milliliters (mL) of water.
- Part A: 200 mg BI 891065 QD: Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered once daily (QD) orally 200 mg of BI 891065, composed of four 50 mg film-coated tablets, with 240 mL of water.
- Part A: 200 mg BI 891065 BID: Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered twice daily (BID) orally 200 mg of BI 891065, composed of four 50 mg film-coated tablets, with 240 mL of water.
Period: Overall Study
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
Started | 3 | 3 | 6
Completed | 0 | 1 | 0
Not Completed | 3 | 2 | 6
Not completed — Clinical disease progression | 0 | 0 | 1
Not completed — Objective disease progression | 3 | 2 | 5

BASELINE CHARACTERISTICS:
Population: The treated set (TS) consisted of all patients who received at least one administration of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (12.1) | 45.7 (7.5) | 54.8 (10.2) | 52.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 8
  Male | 1 | 2 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Patients With Dose Limiting Toxicities (DLTs) in the MTD Evaluation Period
Description: Any of the following adverse events (AEs) were classified as DLTs:
  Haematologic toxicities:
  * Any Grade 5 toxicity.
  * Neutropenia ≥ Grade 4 lasting for >7 days.
  * Febrile neutropenia of any duration (absolute neutrophil count (ANC) <1.0 X 10^9 cells/Liter (L) and fever ≥38.5°Celsius (C)).
  * Neutropenia ≥ Grade 3 with documented infection.
  * Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia with bleeding.
  * Thrombocytopenia of any Grade which requires platelet transfusions.
  * Grade 4 anaemia unexplained by underlying disease.
  * Anaemia of any Grade which requires blood transfusions.
  Non-haematological toxicities:
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times upper level of normal (ULN) and concurrent total bilirubin >2 times ULN without initial findings of cholestasis.
  * ≥Grade 4 AST or ALT of any duration.
  * Any ≥Grade 3 non-haematologic toxicity some exceptions as defined in the protocol.
Time Frame: First treatment cycle, 21 days from first administration of BI 891065.
Population: The MTD evaluation set included all patients who were documented to have received at least one dose of trial medication and were considered evaluable for MTD evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
Number analyzed (Participants) | 3 | 3 | 6
Participants | 1 | 0 | 2
Statistical Analysis 1: Comparison: Part A: 100 mg BI 891065 QD; Probability of DLT rate was determined using a Bayesian 2-parameter logistic regression model with overdose control; Test type: Other; Bayesian logistic regression model; Probability of DLT rate in [0.16,0.33) = 0.172
Statistical Analysis 2: Comparison: Part A: 100 mg BI 891065 QD; Probability of DLT rate was determined using a Bayesian 2-parameter logistic regression model with overdose control; Test type: Other; Probability of DLT rate in [0.33, 1.00] = 0.01
Statistical Analysis 3: Comparison: Part A: 200 mg BI 891065 QD; Probability of DLT rate was determined using a Bayesian 2-parameter logistic regression model with overdose control; Test type: Other; Probabilty of DLT rate in [0.16, 0.33) = 0.362
Statistical Analysis 4: Comparison: Part A: 200 mg BI 891065 QD; Probability of DLT rate was determined using a Bayesian 2-parameter logistic regression model with overdose control; Test type: Other; Probability of DLT rate in [0.33, 1.00] = 0.046
Statistical Analysis 5: Comparison: Part A: 200 mg BI 891065 BID; Probability of DLT rate was determined using a Bayesian 2-parameter logistic regression model with overdose control. The 200 mg BI 891065 BID dose was modelled as equivalent to a 300 mg QD dose in terms of dose-toxicity relationship; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.478
Statistical Analysis 6: Comparison: Part A: 200 mg BI 891065 BID; [analysis description as in outcome 1, analysis 5]; Test type: Other; Probability of DLT rate in [0.33, 1.00] = 0.118

2. Primary Outcome: Part A: Maximum Tolerated Dose (MTD) of BI 891065
Description: Maximum tolerated dose (MTD) of BI 891065 in the Part A of the trial is reported.
  MTD was defined as the highest dose with less than 25% risk of the true DLT rate being equal or above 33% during the MTD evaluation period.
Time Frame: First treatment cycle, 21 days from first administration of BI 891065.
Population: as for outcome 1
Measure: Number; unit: milligram
Groups:
- Part A: BI 891065 All Patients: BI 891065 all patients
Arm/Group | Part A: BI 891065 All Patients
Number analyzed (Participants) | 12
milligram | NA — MTD was not reached during the Part A of the trial because the MTD criteria were not fulfilled for the investigated doses of 100 mg BI 891065 QD, 200 mg BI 891065 QD, and 200 mg BI 891065 BID.

3. Primary Outcome: Part A: Number of Patients With Dose Limiting Toxicities (DLTs) During the Treatment Period
Description: as for outcome 1
Time Frame: From first administration of BI 891065 until the last administration + 30 days of residual effect period, up to 1164 days.
Population: The treated set (TS) consisted of all patients who received at least one administration of trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
Number analyzed (Participants) | 3 | 3 | 6
Participants | 1 | 0 | 2

4. Secondary Outcome: Maximum Measured Concentration in Plasma of BI 891065 After Administration of the First Dose (Cmax)
Description: Maximum measured concentration in plasma of BI 891065 after administration of the first dose (Cmax) is reported.
Time Frame: Within 5 minutes before and 0.5 hours (h), 1h, 2h, 3h, 5h, 6h, 7h, 8h, 10h, 24h, 36h and 48h after first BI 891065 administration.
Population: The pharmacokinetic parameter set (PKS) consisted of all patients in the TS who had at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetic (PK) or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
Number analyzed (Participants) | 3 | 3 | 6
nanomole/Liter | 445 (8.10) | 761 (48.3) | 1270 (45.6)

5. Secondary Outcome: Part A: Maximum Measured Concentration in Plasma of BI 891065 at Steady State (Cmax,ss)
Description: Maximum measured concentration in plasma of BI 891065 at steady state (Cmax,ss) is reported.
Time Frame: Within 5 minutes before and 0.5 hours (h), 1h, 2h, 3h, 5h, 6h, 7h, 8h, 10h and 24 h after drug administration of BI 891065 on Day 15 of Cycle 1.
Population: The pharmacokinetic parameter set (PKS) consisted of all patients in the TS who had at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetic (PK) or due to PK non-evaluability.
  Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
Number analyzed (Participants) | 2 | 3 | 4
nanomole/Liter (nmol/L) | 996 (16.7) | 1370 (15.8) | 4630 (65.6)

6. Secondary Outcome: Part A: Area Under the Concentration-time Curve of BI 891065 in Plasma 24 Hours After Administration of the First Dose (AUC0-24)
Description: Area under the concentration-time curve of BI 891065 in plasma 24 hours after administration of the first dose (AUC0-24) is reported.
Time Frame: Within 5 minutes before and 0.5 hours (h), 1h, 2h, 3h, 5h, 6h, 7h, 8h, 10h and 24h after first administration of BI 891065 on Day 1 of Cycle 1.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanmole/Liter (h*nmol/L)
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
Number analyzed (Participants) | 3 | 3 | 6
hours*nanmole/Liter (h*nmol/L) | 5090 (1.29) | 9410 (52.1) | 15500 (34.6)

7. Secondary Outcome: Part A: Area Under the Concentration-time Curve of BI 891065 in Plasma Over a Uniform Dosing Interval τ at Steady State (AUCτ,ss)
Description: Area under the concentration-time curve of BI 891065 in plasma over a uniform dosing interval τ at steady state (AUCτ,ss) is reported. τ=24 hours (h) for the once daily dosing arms and τ=12 h for the twice daily dosing arm.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours *nanomole/Liter (h*nmol/L)
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
Number analyzed (Participants) | 2 | 3 | 4
hours *nanomole/Liter (h*nmol/L) | 11500 (8.21) | 20500 (15.1) | 47200 (64.8)

ADVERSE EVENTS:
Time Frame: From first administration of BI 891065 until the last administration + 30 days of residual effect period, up to 1164 days.
Description: The treated set (TS) consisted of all patients who received at least one administration of trial medication.
Arm/Group | Part A: 100 mg BI 891065 QD | Part A: 200 mg BI 891065 QD | Part A: 200 mg BI 891065 BID
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 100 mg BI 891065 QD (N=3) | Part A: 200 mg BI 891065 QD (N=3) | Part A: 200 mg BI 891065 BID (N=6)
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 100 mg BI 891065 QD (N=3) | Part A: 200 mg BI 891065 QD (N=3) | Part A: 200 mg BI 891065 BID (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT04138823/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT04138823/SAP_001.pdf